CLINICAL TRIAL: NCT00953745
Title: Dopaminergic Effects of Adjunctive Aripiprazole on the Brain in Treatment-Resistant Depression: A Raclopride/F-DOPA Positron Emission Tomography and Functional MRI Study
Brief Title: Dopaminergic Effects of Adjunctive Aripiprazole on the Brain in Treatment-Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201101790-2
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Neuroimaging; Aripiprazole; Mood disorder; PET Scan; fMRI
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mood Disorders | interventions — Escitalopram; Aripiprazole

STUDY DESIGN:
Intervention Model Description: This study is designed to help understand the mechanism of action of aripiprazole in MDD augmentation. Subjects will undergo exposure to en an existing antidepressant (Lexapro 10-20mg) for 10 weeks; subjects failing to completely respond to the monotherapy antidepressant treatment will receive augmentation with aripiprazole for six weeks. We have included two placebo phases to the study in which the subjects received one placebo along with the Lexapro for the first 6 weeks and a second placebo along with Lexapro for the next two weeks (weeks 7 and 8). This double placebo design is to ensure that subjects receiving aripiprazole augmentation have a legitimate response (non-placebo) to the aripiprazole augmentation. Since the N of this study is small and a small % of patients with placebo response could skew the imaging data significantly, the use of a double placebo prior to the start of the true aripiprazole augmentation should reduce or eliminate a placebo response.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depressed Participants (Active Comparator): Subjects with treatment-resistant depression (TRD) will be administered the Hamilton Depression Rating Scale (HAM-D 17) for entry and will receive escitalopram combined with an adjunctive placebo capsule for 8 weeks.
  Subjects who fail to respond will continue to receive escitalopram and additionally change to receive a placebo tablet resembling the active augmentation agent Aripiprazole (ARP) for 2 weeks.
  Subjects who fail to respond to escitalopram after the 2 phase placebo treatment will enter the ARP augmentation phase of the study and will receive escitalopram augmentation with ARP.
  Subjects will have 3 neuroimaging scans: F-DOPA PET, raclopride PET, and functional MRI conducted after 10 weeks of treatment and repeated after 6 weeks of ARP treatment.
  Interventions: Drug: Escitalopram; Drug: Aripiprazole; Drug: Placebo Capsule; Drug: Placebo Tablet
- Control Participants (No Intervention): Non-depressed, age- and sex-matched subjects without a DSM-IV Axis I diagnosis will serve as controls. They will not receive antidepressant, ARP, or any drug augmentation and will be used as quality control to compare the pre-ARP and post-ARP treatment brain images.

INTERVENTIONS:
Drug: Escitalopram — All subjects will begin on escitalopram and placebo for 8 weeks
  Other Names: Lexapro
  Arms: Depressed Participants
Drug: Aripiprazole — Subjects who fail to respond to Escitalopram will continue on Escitalopram and augment with active Aripiprazole.
  Other Names: Abilify
  Arms: Depressed Participants
Drug: Placebo Capsule — All subjects will begin on escitalopram and placebo capsule for 8 weeks.
  Arms: Depressed Participants
Drug: Placebo Tablet — After 8 weeks, subjects will be given a 2 week supply of escitalopram and placebo tablet.
  Arms: Depressed Participants

SUMMARY:
Aripiprazole has been approved by the FDA for augmenting ineffective/partially effective oral antidepressant therapy in patients suffering from major depression. The mechanism by which this augmentation is achieved is not known. This study has been designed to test the hypothesis that the primary mechanism of action of aripiprazole (ARP) antidepressant augmentation is through the dopaminergic pathway. Two positron emission tomography (PET) scan procedures and a functional magnetic resonance imaging (fMRI) scan will be used to test this hypothesis.

DETAILED DESCRIPTION:
This study is designed to help understand the mechanism of action of ARP in major depressive disorder (MDD) augmentation. Subjects will undergo exposure to an existing antidepressant (Lexapro 10-20mg) for 10 weeks; subjects failing to completely respond to the monotherapy antidepressant treatment will receive augmentation with ARP for six weeks. Two placebo phases are included in which the subjects will receive one placebo along with the Lexapro for the first 6 weeks and a second placebo along with Lexapro for the next two weeks. A baseline brain imaging series (MRI and 2 PET/CT scans) will be obtained at week 10, prior to starting the aripiprazole, on subjects not responding to Lexapro. A second series of images will be obtained at the end of the six weeks of ARP augmentation. The neuroimaging will consist of fMRI, a raclopride PET scan, and a fluoro-dopa PET scan.

Ten normal control subjects will not receive any treatment. They will be age and gender matched to study subjects and undergo one set of scans (fMRI,raclopride and FOPA PET scans) to use as comparison group for quality control on a non-depressed population and not for data analysis.

ELIGIBILITY:
Treatment Group

Inclusion Criteria:

1. Subjects with known history of MDD verified using the Mini International Neuropsychiatric Interview and a Hamilton Depression Rating Scale 17-item score of at least 18
2. Subjects must have failed to respond to one previous adequate dose-duration trial of antidepressant therapy
3. Must complete the MRI screening tool and demonstrate ability to receive an MRI
4. For entry into the ARP augmentation phase the subject must be a non-responder to the escitalopram phase as demonstrated by a MADRS score at week 10, that is not reduced by greater than 50% from baseline.

Exclusion Criteria:

1. Subjects cannot be smokers
2. No significant history of anxiety disorder
3. Cannot be pregnant or lactating and sexually active women of childbearing potential must use a medically accepted means of contraception
4. The following DSM-IV diagnoses are excluded: Organic mental disorder; substance abuse/dependence, including alcohol, active within the last year; schizophrenia, paranoid or delusional disorders; other psychotic disorders; panic disorder; generalized anxiety disorder; obsessive-compulsive disorder, or post-traumatic stress disorder; bipolar disorder; bulimia nervosa; anorexia nervosa
5. Subjects with serious suicidal risks
6. Subjects who have taken any antidepressant medication other than escitalopram within 5 half lives, of the most recent antidepressant taken
7. Subjects involved in any other form of treatment for depression
8. Subjects who have demonstrated any previous inadequate antidepressant response to electroconvulsive therapy (ECT)
9. Subjects who have received ECT for the current depression episode
10. Subjects who have been hospitalized within 4 weeks of the study
11. Subjects who have received treatment with a monoaminoxidase inhibitor within 2 weeks of enrollment
12. Subjects with a known allergy, hypersensitivity, or previous unresponsiveness to aripiprazole or known intolerance to any study medications
13. Subjects with a history of participation in any investigational medication trial in the past month
14. A positive drug screen or substance use disorder in the past 12 months
15. History of any thyroid pathology
16. History of serotonin syndrome or neuroleptic malignant syndrome
17. History of seizure disorder
18. Subjects who have participated in a trial using PET scans in the past 12 months and in any trial in the past 30 days.

Control Group

Inclusion Criteria:

1. Ages 18-55 matched to a study subject
2. Must be a healthy subject with no significant medical history
3. Must complete the MRI screening tool and demonstrate ability to receive an MRI

Exclusion Criteria:

1. Cannot be a smoker
2. Cannot be pregnant or lactating and sexually active women of childbearing potential must use a medically accepted means of contraception
3. Any DSM-IV or II diagnosis as assessed by the MINI
4. Subjects with a positive drug screen or substance use disorder in the past 12 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Depressed Participants: Subjects with treatment-resistant depression (TRD) will receive escitalopram combined with an adjunctive placebo capsule for 8 weeks.
  Subjects who fail to respond will continue to receive escitalopram and additionally change to receive a placebo tablet resembling the active augmentation agent Aripiprazole (ARP) for 2 weeks.
- Control Participants: Non-depressed, age- and sex-matched subjects without a DSM-IV Axis I diagnosis will serve as controls. They will not receive antidepressant, ARP, or any drug augmentation and will be used to compare the pre-ARP and post-ARP treatment brain images to draw conclusions about the pre-treatment state (depression) and post-treatment state (depression responders).
Period: Phase 1: 8 Weeks Escitalopram + Placebo
Arm/Group | Depressed Participants | Control Participants
Started | 37 | 6
Completed | 24 | 6
Not Completed | 13 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Screen failures | 6 | 0
Period: Phase 2: 2 Weeks Escitalopram + Placebo
Arm/Group | Depressed Participants | Control Participants
Started | 18 | 0
Completed | 17 | 0
Not Completed | 1 | 0
Not completed — Pregnancy | 1 | 0
Period: ARP Phase: 6 Weeks Escitalopram + ARP
Arm/Group | Depressed Participants | Control Participants
Started | 17 | 0
Completed | 17 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Depressed Participants: Subjects with treatment-resistant depression (TRD) will receive escitalopram combined with an adjunctive placebo capsule for 8 weeks.
  Subjects who fail to respond will continue to receive escitalopram and additionally change to receive a placebo tablet resembling the active augmentation agent Aripiprazole (ARP) for 2 weeks.
  Subjects who fail to respond to escitalopram after the 2 phase placebo treatment will enter the ARP augmentation phase of the study and will receive escitalopram augmentation with ARP.
  Subjects will have 3 neuroimaging scans: F-DOPA PET, raclopride PET, and functional MRI conducted after 10 weeks of treatment and repeated after 6 weeks of ARP treatment.
- Total: Total of all reporting groups
Arm/Group | Depressed Participants | Control Participants | Total
Number analyzed (Participants) | 37 | 6 | 43
Age, Continuous [Mean (Full Range); unit: years] | 41.69 [19 to 54] | 45.67 [31 to 54] | 42.27 [19 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 5 | 32
  Male | 10 | 1 | 11
Region of Enrollment [Number; unit: participants]
  United States | 37 | 6 | 43

OUTCOME MEASURES:

1. Primary Outcome: Fluorodopa Uptake Values in Brain Images of Aripiprazole Augmentation Responders
Description: A ratio of the image derived radioactivity concentration and the whole body concentration of the injected radioactivity specifically in a cluster within the right medial caudate (see data below).
Time Frame: Week 10 and Week 16 (6 weeks of combined therapy)
Population: The outcome purpose was to examine mechanism of action of aripiprazole in responders versus nonresponders. Control subjects were age and gender matched to study subjects and underwent one set of scans (fMRI, raclopride and FOPA PET scans) for use as a comparison group for quality control on a non-depressed population and not for data analysis.
Measure: Mean (Standard Deviation); unit: FDOPA ratio in the right medial caudate
Groups:
- ARP Responders; ARP Non-Responders: Subjects who fail to respond to escitalopram after the 2 phase placebo treatment will enter the ARP augmentation phase of the study and will receive escitalopram augmentation with ARP. ARP Responders will have had a 50% or greater drop in their MADRS scores from baseline.
  Subjects will have 3 neuroimaging scans: F-DOPA PET, raclopride PET, and functional MRI conducted after 10 weeks of treatment and repeated after 6 weeks of ARP treatment.
Arm/Group | ARP Responders | ARP Non-Responders
Number analyzed (Participants) | 11 | 3
FDOPA ratio in the right medial caudate
  Week 10 | 1.297 (0.176) | 1.363 (0.180)
  Week 16 | 1.333 (0.175) | 1.350 (0.252)
Statistical Analysis 1: Comparison: ARP Responders; A region of increased relative Fluorodopa (FDOPA) uptake in the right medial caudate was anticipated for the aripiprazole augmentation responders over the 6 weeks of augmentation treatment (Weeks 10-16); Test type: Superiority or Other; p = 0.029, t-test, 1 sided — paired t-test thresholded at cluster level significance of p=0.001; family-wise error multiple comparisons corrected

2. Secondary Outcome: Depression Symptom Change on The Montgomery-Åsberg Depression Rating (MADRS) Scale Between ARP Responders and Non-responders.
Description: Montgomery-Åsberg Depression Rating (MADRS) Scale scores compared between the 6 week Aripiprazole augmentation groups (responds vs. non-responders). Total range of the MADRS is 0 to 60, with a score of greater than 34 indicating severe depression, 20-34 indicating moderate depression, 7-19 mild depression, and 0-6 normal or absent of symptoms.
Time Frame: Week 10 and Week 16 (6 weeks of combined therapy)
Population: MADRS score comparison between ARP responders and nonresponders.
Measure: Mean (Standard Deviation); unit: score on the MADRS scale
Groups:
- ARP Responders: Subjects who fail to respond to escitalopram after the 2 phase placebo treatment will enter the ARP augmentation phase of the study and will receive escitalopram augmentation with ARP. ARP Responders will have had a 50% or greater drop in their MADRS scores from baseline.
- ARP Non-Responders: Subjects who fail to respond to escitalopram after the 2 phase placebo treatment will enter the ARP augmentation phase of the study and will receive escitalopram augmentation with ARP. ARP non-responders will not have had a 50% or greater drop in their MADRS scores from baseline.
Arm/Group | ARP Responders | ARP Non-Responders
Number analyzed (Participants) | 11 | 3
score on the MADRS scale
  Week 10 | 27.9 (5.6) | 31.7 (12.7)
  Week 16 | 6.5 (3.0) | 25.3 (5.5)
Statistical Analysis 1: Comparison: ARP Responders; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: ARP Non-Responders; Test type: Superiority or Other; p = 0.366, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Depressed Participants | Control Participants
Serious Adverse Events (participants affected / at risk) | 2/37 | 0/6
Other Adverse Events (participants affected / at risk) | 24/37 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Depressed Participants (N=37) | Control Participants (N=6)
Birth of a baby (deception by subject) (Pregnancy, puerperium and perinatal conditions) | 1/27 (1) | 0 (0) — Subject documented as non pregnant/breast-feeding. Five urine pregnancy tests conducted within 10 weeks prior to the birth of her full term baby; all were negative (subject provided fake urine). Terminated from study upon date of discovery.
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/27 (1) | 0 (0) — Occurred ~4 weeks after start of escitalopram; continued an additional 4 weeks. Admitted noncompliance to use of acceptable birth control method. Terminated from study. Subject reported escitalopram discontinuation and delivery of a healthy baby.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Depressed Participants (N=37) | Control Participants (N=6)
Increased fatigue (Nervous system disorders) | 11 | 0
Nausea (Gastrointestinal disorders) | 7 | 0
Akathisia (Nervous system disorders) | 4 | 0
Insomnia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 0
Increased sweating (Nervous system disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Lightheadedness (Ear and labyrinth disorders) | 2 | 0
Restlessness (Nervous system disorders) | 4 | 0
Decreased libido (Nervous system disorders) | 3 | 0
Vivid dreaming (Nervous system disorders) | 4 | 0
Dizziness (Ear and labyrinth disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes